CLINICAL TRIAL: NCT01707888
Title: VATS Major Lung Resection for Chinese Early-stage Non-small Cell Lung cancer-a Registry Study
Brief Title: VATS Major Lung Resection for Chinese Early-stage Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jun Wang, Principal Investigator, Clinical Professor, Peking University People's Hospital
Other Study IDs: PEKUPH1201
Record Dates: First submitted 2012-10-13; First posted 2012-10-16 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- major lung resection: Patients undergo major lung resection by thoracoscopy/VATS.
  Interventions: Procedure: Thoracoscopy/VATS

INTERVENTIONS:
Procedure: Thoracoscopy/VATS — Patients undergo major lung resection by thoracoscopic surgery or video assisted thoracoscopic surgery.
  Other Names: Minimal invasive surgery

SUMMARY:
Surgery may be the best treatment choice for early stage non-small cell lung cancer. And VATS major lung resection have been preferred as a standard radical procedure for early stage non-small cell lung cancer (NSCLC).This study aim to investigate the outcome of VATS major lung resection for lung cancer as a real-world study in china.

DETAILED DESCRIPTION:
Surgery may be the best treatment choice for early stage non-small cell lung cancer. And VATS major lung resection have been preferred as a standard radical procedure for early stage non-small cell lung cancer (NSCLC).This study aim to investigate the outcome of VATS major lung resection for lung cancer as a real-world study in china.This is a multicenter, prospective study, aimed To evaluate the short-term and long- term outcome of VATS major lung resection for early stage lung cancer. Patients will be followed up every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

Preoperative criteria:

i) non-small cell lung cancer is suspected, ii) clinical stage I/II (3) Intraoperative criteria: i) Histologically confirmed NSCLC, ii) resected by VATS or converted open lobectomy,sleeve lobectomy or pneumonectomy and nodal dissection/sampling.

(4) No prior ipsilateral thoracotomy (prior diagnostic thoracoscopy is allowed).

(5) No prior chemotherapy or radiation therapy for any malignant diseases. (6) Expected postoperative FEV1.0>=800 mL and PaO2>=65 torr. (7) Performance status of 0 or 1. (8) Sufficient organ functions. (9) Written informed consent.

Exclusion Criteria:

1. Active bacterial or fungous infection.
2. Simultaneous or metachronous (within the past 5 years) double cancers.
3. Women during pregnancy or breast-feeding.
4. Interstitial pneumonitis, pulmonary fibrosis, or severe pulmonary emphysema.
5. Psychosis.
6. Systemic steroids medication.
7. Uncontrollable diabetes mellitus.
8. Uncontrollable hypertension.
9. History of severe heart disease, heart failure, myocardial infarction within the past 6 months or attack of angina pectoris within the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinical early stage(I/II) lung cancer
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
morbidity and mortility rate | 3 moths
  perioperative complications and death rates of the group

SECONDARY OUTCOMES:
Disease-free survival | 3y
  To evaluate Disease Free Survival (DFS) of the group.
Rate of loco-regional and systemic recurrence | 3y
  To evaluate the rate of loco-regional and systemic recurrence of the group.
Pulmonary function | 6 months after surgery
  to evaluate the pulmonary function as measured by expiratory flow rate of the group 6 months postoperatively.
Postoperative hospital stay. | 3 months postoperatively
  to evaluate the postoperative hospital stay of the group.
Postoperative drainage duration | 3 months postoperatively
  to evaluate the postoperative drainage duration of the group.
overall survival | 3 months postoperatively
  to evaluate the overall survival rate of the group.
converted rate | 3 months
  the rate of converted thoracotomy

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, MD, Study Chair — Peking University People's Hospital; Fan Yang, MD, Study Director — Peking University People's Hospital; Zhao Xi Sui, MD, Study Director — Peking University People's Hospital
Locations (6):
- China (6):
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chao-Yang Hospital, Beijing, Beijing Municipality
  - Beijing Haidian Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing
  - Peking university people's hospital, Beijing